CLINICAL TRIAL: NCT05274776
Title: Safely Reduce Newborn Antibiotic Exposure With the Early-onset Sepsis Calculator: a Cluster Randomized Study (EOS Calculator RCT)
Brief Title: Safely Reduce Newborn Antibiotic Exposure With the Early-onset Sepsis Calculator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: prof. dr. Frans B. Plötz (Other)
Collaborators: Dutch Society of Pediatrics (Unknown); Zorgevaluatie Nederland (Unknown); Care4Neo (Unknown); everywhereIM (Unknown)
Responsible Party: Sponsor-Investigator, prof. dr. Frans B. Plötz, Professor of Pediatric Health Care Evaluation, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL78203.018.21
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Early-Onset Sepsis, Neonatal; EOS
Keywords: early-onset sepsis; neonatal; EOS calculator
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: A prospective, cluster-randomized trial will be conducted; five hospitals will be randomized to NVK guidelines use, five hospitals will be randomized to EOS calculator use. After randomization, the assigned protocol is considered standard care for newborns with suspected EOS within 0-24 hours after birth during the study period in that hospital. This means that the NVK guidelines or the EOS calculator (depending on randomization) will be used for all newborns at risk for EOS (within 0-24 hours after birth) in the assigned hospital, independent of study participation. It is noteworthy that attending physicians have the option to choose for clinical management according to another protocol instead of the assigned protocol.
Masking Description: Hospitals nor physicians are blinded for the assigned study protocol. Since the assigned protocol is considered standard care for newborns with suspected EOS within 0-24 hours after birth during the study period in that hospital, independent of study participation, parents of participants are not blinded as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVK Guidelines (No Intervention): The NVK guidelines use 8 maternal and 15 neonatal risk factors, each categorized as either red flag or non-red flag. These criteria guide clinicians on the management in case of suspected EOS. Briefly, antibiotic treatment is recommended if at least one red flag and, or, two or more non-red flags are present. An observation period of at least 12 hours is recommended if one non-red flag is present. Antibiotics are recommended when an infection is suspected during this observation. Newborns without EOS risk factors, with a good clinical condition, and a gestational age of more than 36 weeks will be discharged. If the guidelines recommend an observation period, the newborn with a good clinical condition is discharged after repeating physical examination. In case antibiotic treatment is started, discharge depends on the duration of treatment and the clinical course. At discharge, parents are instructed to call the hospital in case of signs of infection within the first 14 days of life.
- EOS Calculator (Experimental): Using the EOS calculator application between 0-24 hours after birth, maternal EOS risk factors combined with the physical examination of the newborn are used to assign a risk category and accompanying clinical recommendation based on estimated EOS incidence for each newborn at-risk for an infection. The EOS calculator results are used to guide clinical management on performing either a diagnostic work-up and start of antibiotics for (suspected) EOS, or a conservative approach with routine controls of vital parameters every 3 hours. In case of routine controls, re-evaluation of physical appearance by a pediatric resident or pediatrician will take place within 24 hours postpartum. Newborns will be observed for at least 24 hours. In case antibiotics are started, the need for further treatment is depending on blood culture results, infection parameters, and clinical condition of the newborn. Discontinuation of antibiotics and discharge is at the discretion of the treating physician.
  Interventions: Device: EOS calculator

INTERVENTIONS:
Device: EOS calculator — For this study the EOS calculator was developed as a mobile application (by everywhereIM), including CE marking. It is concerned a medical device for health care professionals.
  Other Names: early-onset sepsis calculator; neonatal early-onset sepsis calculator; sepsis risk calculator (SRC); newborn sepsis calculator; neonatal EOS calculator
  Arms: EOS Calculator

SUMMARY:
Newborns are at risk for early-onset sepsis (EOS), which occurs within 72 hours after birth. The incidence of proven EOS is 0.5-2.0 per 1000 live births. The annual birth rate in the Netherlands is around 170.000, consequently the number of EOS cases varies between 85 to 340. However, about 5%, thus 8500, of late preterm and term newborns receive empiric antibiotic therapy in compliance with the current Dutch guideline. An alternative is the CE certified EOS calculator application, which calculates an individual EOS risk with treatment advice. In this prospective cluster-randomized multicenter trial the current Dutch guideline will be compared with the EOS calculator in newborns at risk for EOS.

The primary objectives of this study are:

1. To investigate whether the use of the EOS calculator reduces antibiotic exposure in newborns with suspected EOS in the first 24 hours after birth.
2. To investigate the presence of one or more of the following four predefined safety criteria, namely 1) the need for any respiratory support, and/or 2) the need for an intravascular fluid bolus for hemodynamic instability due to sepsis, and/or 3) referral to a Neonatal Intensive Care Unit for sepsis treatment, and/or 4) proven EOS.

Secondary objectives of the study are:

1. To investigate if the use of the EOS calculator decreases the total duration of antibiotic therapy in newborns with suspected EOS.
2. To investigate if the use of the EOS calculator decreases the percentage of antibiotic therapy started for suspected and, or proven EOS if symptoms started between 24-72 hours after birth.
3. To study the impact of (suspected) EOS on parents/guardians.

DETAILED DESCRIPTION:
Suspicion of EOS is often based on risk factors and nonspecific clinical symptoms, such as maternal fever during labor or rapid breathing in the newborn. The combination of the difficulty to recognize EOS in time and the risk of serious consequences of EOS not treated timely has resulted in a low threshold for the start of empirical antibiotic therapy. This has led to significant overtreatment.

The current standard of care in the Netherlands is the Dutch Society of the Nederlands (NVK) guideline "Prevention and treatment of early-onset neonatal infections", which is an adaptation of the 2012 version of the National Institute for Health and Care Excellence (NICE) guideline "Antibiotics for early-onset neonatal infection: antibiotics for the prevention and treatment of early-onset neonatal infection". The NVK guideline uses risk factors and symptoms to categorically indicate which newborns need antibiotic therapy. Evaluating its use in 9 Dutch hospitals, limited adherence was found, especially when antibiotics were recommended by the guideline but withheld by the clinicians. This limited adherence indicates that it is desirable to amend the current guideline or to investigate the use of an alternative method.

A new method for determining which newborns need antibiotic therapy is the "EOS calculator". Developed in the United States, this method uses a combination of detailed information about 5 maternal risk factors and the presence of clinical neonatal symptoms to calculate an individual EOS risk and treatment advice.

For the Dutch situation, equipoise between the current NVK guideline and the EOS calculator can be established given balance of risk for both over- and undertreatment of EOS for both strategies. A large body of evidence now supports the safety of the EOS calculator approach, but validation outside of the North-American setting is limited, especially for safety outcomes.

A prospective cluster-randomized Dutch validation study of the EOS calculator is needed before implementation because of the following reasons:

1. Multicenter validation of actual EOS calculator use has not been performed in the Netherlands.
2. To date, no randomized prospective study of EOS calculator use with safety as an outcome measure has been performed. Specifically, there are no studies that take into account the potential effects of a treatment delay due to EOS calculator use. This especially holds true for cases that are clinically suspect for EOS, but not culture-confirmed.

ELIGIBILITY:
Inclusion Criteria:

* postmenstrual age of 34 weeks or more;
* age between 0-24 hours;
* at least one EOS risk factor or clinical sign of infection (suspected of EOS) present within the first 24 hours of life;
* parental/guardian consent.

Exclusion Criteria:

* major congenital anomalies;
* language barrier (lack of effective communication or whenever it hinders understanding).

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1830 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Co-primary superiority outcome: antibiotic therapy started within 24 hours after birth | 0-24 hours after birth
  The proportion of patients that started antibiotic therapy for suspected and, or proven EOS in the first 24 hours after birth.
First co-primary non-inferiority outcome (safety): proportion of patients with respiratory support | 0-14 days after birth
  A composite non-inferiority outcome regarding the presence of one or more of the following four predefined safety criteria, namely 1) the need for any respiratory support, and/or 2) the need for an intravascular fluid bolus for hemodynamic instability due to sepsis, and/or 3) referral to a Neonatal Intensive Care Unit (NICU) for sepsis treatment, and/or 4) proven EOS.
  - Respiratory support is defined as any form of respiratory support (invasive ventilation, continuous positive airway pressure (CPAP), high flow nasal cannula (HFNC), low flow oxygen) during the first week of life.
Second co-primary non-inferiority outcome (safety): proportion of patients with hemodynamic support | 0-14 days after birth
  - Intravascular fluid bolus is defined as the intravenous administration of a fluid bolus of 10ml/kg within 15-30 minutes. It is the first step in the treatment of hemodynamically unstable newborns due to sepsis.
Third co-primary non-inferiority outcome (safety): proportion of patients referred to a NICU for sepsis treatment | 0-14 days after birth
Fourth co-primary non-inferiority outcome (safety): proportion of patients with proven EOS | 0-14 days after birth
  - Proven EOS is defined as a blood or cerebrospinal fluid (CSF) culture obtained within 72 hours after birth growing a pathogenic bacterial species.

SECONDARY OUTCOMES:
Duration of antibiotic therapy | 0-14 days after birth
  The total duration of antibiotic therapy: date and time of first administration of intravenous antibiotic therapy, and date and time of the last administration of intravenous antibiotic therapy.
Antibiotic therapy started between 24-72 hours after birth | 24-72 hours after birth
  The proportion of antibiotic therapy started for suspected and, or proven EOS if symptoms started between 24-72 hours after birth.
Questionnaire: quality of life | 14-28 days after birth
  To get an impression of the impact of (suspected) early-onset sepsis on the quality of life (QoL) of both parents/guardians and their child, parents/guardians will be asked to fill in a questionnaire on day 14 after birth. The first part collects information on medical factors after hospitalization (side effects, number of medical visits, readmission, and medication use) and basic needs of the newborn (sleep quality of the patient, (breast)feeding success rate). The second part addresses the subjective parental/guardian evaluation of the impact of newborns' admission, and parental/guardian projection of future QoL of their newborn. Statements with six possible answers will be used: 'not at all, a little, on average, more than average, a lot, not applicable' or 'poor, fair, good, very good, excellent, not applicable'. Participants will not score on a numbered scale but tick the answer (in text) that apply best. The last part of the questionnaire collects demographic data.

CONTACTS AND LOCATIONS:
Overall Officials: Frans B. Plötz, MD, PhD, Principal Investigator — Amsterdam UMC, Tergooi Ziekenhuizen; Niek B. Achten, MD, PhD, Study Director — Erasmus Medical Center; Bo M. van der Weijden, MD, Study Director — Amsterdam UMC, Tergooi Ziekenhuizen
Locations (10):
- Netherlands (10):
  - Northwest Clinics, Alkmaar
  - FlevoHospital, Almere Stad
  - Amstelland Hospital, Amstelveen
  - OLVG, Amsterdam
  - Martini Hospital, Groningen
  - Spaarne Hospital, Haarlem
  - Dijklander Hospital, Hoorn
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Máxima Medical Center, Veldhoven
  - Zaans Medical Centre, Zaandam

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request through a repository and shared after consent of the principal investigator.

REFERENCES:
- [Background] Shane AL, Sanchez PJ, Stoll BJ. Neonatal sepsis. Lancet. 2017 Oct 14;390(10104):1770-1780. doi: 10.1016/S0140-6736(17)31002-4. Epub 2017 Apr 20. PMID 28434651
- [Background] Sagori Mukhopadhyay, Karen M. Puopolo; Neonatal Early-Onset Sepsis: Epidemiology and Risk Assessment. Neoreviews April 2015; 16 (4): e221-e230.
- [Background] Simonsen KA, Anderson-Berry AL, Delair SF, Davies HD. Early-onset neonatal sepsis. Clin Microbiol Rev. 2014 Jan;27(1):21-47. doi: 10.1128/CMR.00031-13. PMID 24396135
- [Background] Klingenberg C, Kornelisse RF, Buonocore G, Maier RF, Stocker M. Culture-Negative Early-Onset Neonatal Sepsis - At the Crossroad Between Efficient Sepsis Care and Antimicrobial Stewardship. Front Pediatr. 2018 Oct 9;6:285. doi: 10.3389/fped.2018.00285. eCollection 2018. PMID 30356671
- [Background] Cantey JB, Wozniak PS, Pruszynski JE, Sanchez PJ. Reducing unnecessary antibiotic use in the neonatal intensive care unit (SCOUT): a prospective interrupted time-series study. Lancet Infect Dis. 2016 Oct;16(10):1178-1184. doi: 10.1016/S1473-3099(16)30205-5. Epub 2016 Jul 22. PMID 27452782
- [Background] Korpela K, Zijlmans MA, Kuitunen M, Kukkonen K, Savilahti E, Salonen A, de Weerth C, de Vos WM. Childhood BMI in relation to microbiota in infancy and lifetime antibiotic use. Microbiome. 2017 Mar 3;5(1):26. doi: 10.1186/s40168-017-0245-y. PMID 28253911
- [Background] Low JSY, Soh SE, Lee YK, Kwek KYC, Holbrook JD, Van der Beek EM, Shek LP, Goh AEN, Teoh OH, Godfrey KM, Chong YS, Knol J, Lay C. Ratio of Klebsiella/Bifidobacterium in early life correlates with later development of paediatric allergy. Benef Microbes. 2017 Oct 13;8(5):681-695. doi: 10.3920/BM2017.0020. Epub 2017 Oct 12. PMID 29022383
- [Background] NVOG (Nederlandse Vereniging voor Obstetrie en Gynaecologie), NVK (Nederlandse Vereniging Kindergeneeskunde). Preventie en behandeling van early-onset neonatale infecties (Adaptatie van de NICE-richtlijn). 2017 p. 1-94.
- [Background] Neonatal infection: antibiotics for prevention and treatment. London: National Institute for Health and Care Excellence (NICE); 2024 Mar 19. Available from http://www.ncbi.nlm.nih.gov/books/NBK571222/ PMID 34133110
- [Background] van der Weijden BM, Achten NB, Bekhof J, Evers EE, Berk M, Kamps AWA, Rijpert M, Ten Tusscher GW, van Houten MA, Plotz FB. Multicentre study found that adherence to national antibiotic recommendations for neonatal early-onset sepsis was low. Acta Paediatr. 2021 Mar;110(3):791-798. doi: 10.1111/apa.15488. Epub 2020 Aug 10. PMID 32686180
- [Background] Escobar GJ, Puopolo KM, Wi S, Turk BJ, Kuzniewicz MW, Walsh EM, Newman TB, Zupancic J, Lieberman E, Draper D. Stratification of risk of early-onset sepsis in newborns >/= 34 weeks' gestation. Pediatrics. 2014 Jan;133(1):30-6. doi: 10.1542/peds.2013-1689. Epub 2013 Dec 23. PMID 24366992
- [Background] Puopolo KM, Draper D, Wi S, Newman TB, Zupancic J, Lieberman E, Smith M, Escobar GJ. Estimating the probability of neonatal early-onset infection on the basis of maternal risk factors. Pediatrics. 2011 Nov;128(5):e1155-63. doi: 10.1542/peds.2010-3464. Epub 2011 Oct 24. PMID 22025590
- [Background] Kuzniewicz MW, Puopolo KM, Fischer A, Walsh EM, Li S, Newman TB, Kipnis P, Escobar GJ. A Quantitative, Risk-Based Approach to the Management of Neonatal Early-Onset Sepsis. JAMA Pediatr. 2017 Apr 1;171(4):365-371. doi: 10.1001/jamapediatrics.2016.4678. PMID 28241253
- [Background] Achten NB, Klingenberg C, Benitz WE, Stocker M, Schlapbach LJ, Giannoni E, Bokelaar R, Driessen GJA, Brodin P, Uthaya S, van Rossum AMC, Plotz FB. Association of Use of the Neonatal Early-Onset Sepsis Calculator With Reduction in Antibiotic Therapy and Safety: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Nov 1;173(11):1032-1040. doi: 10.1001/jamapediatrics.2019.2825. PMID 31479103
- [Background] Achten NB, Dorigo-Zetsma JW, van der Linden PD, van Brakel M, Plotz FB. Sepsis calculator implementation reduces empiric antibiotics for suspected early-onset sepsis. Eur J Pediatr. 2018 May;177(5):741-746. doi: 10.1007/s00431-018-3113-2. Epub 2018 Feb 18. PMID 29455368
- [Background] van der Weijden BM, Achten NB, Bekhof J, Evers EE, van Dongen O, Rijpert M, Kamps AWA, Ten Tusscher GW, van Houten MA, Plotz FB. Neonatal early-onset sepsis calculator recommended significantly less empiric antibiotic treatment than national guidelines. Acta Paediatr. 2020 Dec;109(12):2549-2551. doi: 10.1111/apa.15391. Epub 2020 Jun 17. No abstract available. PMID 32497338
- [Background] Achten NB, Klingenberg C, Plotz FB. Neonatal Early-Onset Sepsis Calculator and Antibiotic Therapy-Reply. JAMA Pediatr. 2020 May 1;174(5):508-509. doi: 10.1001/jamapediatrics.2019.6269. No abstract available. PMID 32150235
- [Background] Kerste M, Corver J, Sonnevelt MC, van Brakel M, van der Linden PD, M Braams-Lisman BA, Plotz FB. Application of sepsis calculator in newborns with suspected infection. J Matern Fetal Neonatal Med. 2016 Dec;29(23):3860-5. doi: 10.3109/14767058.2016.1149563. Epub 2016 Mar 7. PMID 26948457
- [Background] Achten, N. B., Zonneveld, R., Tromp, E., & Plotz, F. B. (2017). Association between sepsis calculator and infection parameters for newborns with suspected early onset sepsis. Journal of clinical neonatology, 6(3), 159-162.
- [Background] Achten NB, Visser DH, Tromp E, Groot W, van Goudoever JB, Plotz FB. Early onset sepsis calculator implementation is associated with reduced healthcare utilization and financial costs in late preterm and term newborns. Eur J Pediatr. 2020 May;179(5):727-734. doi: 10.1007/s00431-019-03510-9. Epub 2020 Jan 2. PMID 31897840
- [Background] Achten NB, Dorigo-Zetsma JW, van Rossum AMC, Oostenbrink R, Plotz FB. Risk-based maternal group B Streptococcus screening strategy is compatible with the implementation of neonatal early-onset sepsis calculator. Clin Exp Pediatr. 2020 Oct;63(10):406-410. doi: 10.3345/cep.2020.00094. Epub 2020 Apr 16. PMID 32299178
- [Background] Benitz WE, Achten NB. Finding a role for the neonatal early-onset sepsis risk calculator. EClinicalMedicine. 2020 Jan 26;19:100255. doi: 10.1016/j.eclinm.2019.100255. eCollection 2020 Feb. No abstract available. PMID 32140673
- [Background] Benitz WE, Achten NB. Technical assessment of the neonatal early-onset sepsis risk calculator. Lancet Infect Dis. 2021 May;21(5):e134-e140. doi: 10.1016/S1473-3099(20)30490-4. Epub 2020 Oct 29. PMID 33129425
- [Background] Achten NB, Plotz FB, Klingenberg C, Stocker M, Bokelaar R, Bijlsma M, Giannoni E, van Rossum AMC, Benitz WE. Stratification of Culture-Proven Early-Onset Sepsis Cases by the Neonatal Early-Onset Sepsis Calculator: An Individual Patient Data Meta-Analysis. J Pediatr. 2021 Jul;234:77-84.e8. doi: 10.1016/j.jpeds.2021.01.065. Epub 2021 Feb 3. PMID 33545190
- [Background] Counsilman CE, Heeger LE, Tan R, Bekker V, Zwaginga JJ, Te Pas AB, Lopriore E. Iatrogenic blood loss in extreme preterm infants due to frequent laboratory tests and procedures. J Matern Fetal Neonatal Med. 2021 Aug;34(16):2660-2665. doi: 10.1080/14767058.2019.1670800. Epub 2019 Oct 6. PMID 31588840
- [Background] Kuzniewicz MW, Walsh EM, Li S, Fischer A, Escobar GJ. Development and Implementation of an Early-Onset Sepsis Calculator to Guide Antibiotic Management in Late Preterm and Term Neonates. Jt Comm J Qual Patient Saf. 2016 May;42(5):232-9. doi: 10.1016/s1553-7250(16)42030-1. No abstract available. PMID 27066927
- [Background] Keij FM, Kornelisse RF, Hartwig NG, Mauff K, Poley MJ, Allegaert K, Reiss IKM, Tramper-Stranders GA. RAIN study: a protocol for a randomised controlled trial evaluating efficacy, safety and cost-effectiveness of intravenous-to-oral antibiotic switch therapy in neonates with a probable bacterial infection. BMJ Open. 2019 Jul 9;9(7):e026688. doi: 10.1136/bmjopen-2018-026688. PMID 31289068
- [Background] Ferrand A, Gorgos A, Ali N, Payot A. Resilience Rather than Medical Factors: How Parents Predict Quality of Life of Their Sick Newborn. J Pediatr. 2018 Sep;200:64-70.e5. doi: 10.1016/j.jpeds.2018.05.025. Epub 2018 Jun 27. PMID 29958673
- [Background] NFU (Dutch Federation of University Medical Centers). Richtlijn Kwaliteitsborging Mensgebonden Onderzoek 2020. 2020.
- [Background] Cotten CM. Adverse consequences of neonatal antibiotic exposure. Curr Opin Pediatr. 2016 Apr;28(2):141-9. doi: 10.1097/MOP.0000000000000338. PMID 26886785
- [Background] Zven SE, Susi A, Mitre E, Nylund CM. Association Between Use of Multiple Classes of Antibiotic in Infancy and Allergic Disease in Childhood. JAMA Pediatr. 2020 Feb 1;174(2):199-200. doi: 10.1001/jamapediatrics.2019.4794. PMID 31860016
- [Background] van Herk W, Stocker M, van Rossum AM. Recognising early onset neonatal sepsis: an essential step in appropriate antimicrobial use. J Infect. 2016 Jul 5;72 Suppl:S77-82. doi: 10.1016/j.jinf.2016.04.026. Epub 2016 May 21. PMID 27222092
- [Background] National Institute for Health and Care Excellence. Neonatal infection (early onset): Antibiotics for prevention and treatment. Clinical Guideline. 2012
- [Derived] van der Weijden BM, Janssen SWCM, van der Weide MC, Cornelisse-van Vugt RJPM, Ten Tusscher GW, Lutterman CAM, Kamps AWA, Lorente Flores CM, Hol J, van Laerhoven H, Rijpert M, Oeij NA, Schiering IAM, Obermann-Borst SA, Visser DH, van Leeuwen LM, Kornelisse RF, van Rossum AMC, Bijlsma MW, Plotz FB, Achten NB. Safety and effectiveness of the early-onset sepsis calculator to reduce antibiotic exposure in at-risk newborns: a cluster-randomised controlled trial. EClinicalMedicine. 2025 Aug 12;87:103419. doi: 10.1016/j.eclinm.2025.103419. eCollection 2025 Sep. PMID 40831464
- [Derived] van der Weijden BM, van der Weide MC, Plotz FB, Achten NB. Evaluating safety and effectiveness of the early-onset sepsis calculator to reduce antibiotic exposure in Dutch at-risk newborns: a protocol for a cluster randomised controlled trial. BMJ Open. 2023 Feb 14;13(2):e069253. doi: 10.1136/bmjopen-2022-069253. PMID 36787971
- See also: Webpage of Zorgevaluatie Nederland, where everybody can find all study-related information, documents and progress. — https://zorgevaluatienederland.nl/evaluations/eos-calculator-rct